CLINICAL TRIAL: NCT06242951
Title: Cardiopulmonary Fitness in Children With Cystic Fibrosis Compared to Healthy Children
Acronym: VOmuco
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-MTP_2023_01_202201310
Record Dates: First submitted 2023-12-22; First posted 2024-02-05 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis in Children
Keywords: VO2 max; cardiopulmonary exercise test; physical fitness; pediatrics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: Patients with cystic fibrosis
  Interventions: Diagnostic Test: VO2 max assessment
- Control
  Interventions: Diagnostic Test: VO2 max assessment

INTERVENTIONS:
Diagnostic Test: VO2 max assessment — Measurement of the maximum oxygen consumption (VO2max) by a cardiopulmonary exercise test (CPET)

SUMMARY:
Cystic fibrosis is the most common severe genetic disease with autosomal recessive transmission in the Caucasian population.

Its prognosis has improved considerably since the creation of Cystic Fibrosis centers (CF centers) and the improvement of symptomatic management (nutrition, antibiotic therapy, transplantation, etc.). Thus, the median survival rate is now 46 years, whereas it was 5 years in 1963.

The current challenges for cystic fibrosis patients are therefore twofold:

to continue to improve their survival, and to improve their quality of life (QoL) to promote "healthy ageing" with this pathology that begins in childhood.

In 1980, the World Health Organization (WHO) stated that functional capacity explorations best reflected the impact of chronic disease on health-related quality of life. Impairment of physical activity is common to chronic diseases, as in cystic fibrosis, where respiratory impairment and denutrition have been shown to contribute to reduced exercise tolerance and increased dyspnoea.

Measurement of the maximum oxygen consumption (VO2max) by a cardiopulmonary exercise test (CPET) is regarded as the gold standard exercise test in the measurement of aerobic exercise capacity.

In 2005 Pianosi et al. found that for children with cystic fibrosis, the rate of decline of VO2max measured by CPET was predictive of poorer quality of life.

Continuing to study the determinants associated with impaired aerobic fitness in cystic fibrosis offers the hope of considering appropriate therapies to further improve the quality of life of these patients.

In recent years, the arrival and widespread use of CFTR protein modulators in children has been a real turning point and makes it possible to envisage a drastic change in the history of this disease and its prognosis in the long term.

Thus, in this study, the investigators aimed to assess the aerobic fitness, assessed by a CPET, of children with cystic fibrosis, and to compare the results with healthy controls. Secondly, investigators wanted to identify the predictive factors of VO2max in children with cystic fibrosis.

DETAILED DESCRIPTION:
This retrospective study was carried out from November 2010 to September 2015 for control children (already published PubMed Identifier (PMID): 29170358) : and July 2018 to December 2019 for cystic fibrosis children.

CPET were performed in the paediatric CPET laboratory of Montpellier University Hospital, France.

Children aged 7 to 17 years old were recruited. Two groups were identified: children with cystic fibrosis and healthy control children.

1. The cystic fibrosis group consisted of children followed up every three months in the cystic fibrosis center of Montpellier University and referred to our paediatrician CPET laboratory in 2019 in the framework of an annual check-up. For the few patients who did not have a CPET in 2019, investigators included those who passed a CPET between July and December 2018. From patients' interviews, the absence of any physical activity, apart from physical education at school, was indicative of sedentary lifestyle.

   Investigators also collected anthropometric data, radiological findings, CF-related markers of disease severity including cystic fibrosis transmembrane conductance regulator (CFTR) genotype, microbiological infection, pancreatic insufficiency, cystic fibrosis-related diabetes (CFRD), and treatment including modulator data.
2. As in our previous similar CPET controlled paediatric studies, the control group consisted of children referred for non-severe functional symptoms linked to exercise (murmur, palpitation or dyspnoea) or for medical sports certificate. These children were classified as controls after a completely normal check-up, including physical examination, ECG, echocardiography and spirometry. Children with any chronic disease, medical condition (cardiac, neurologic, respiratory, muscular or renal), or medical treatment, and those requiring any further specialised medical consultation were not eligible.

CPET procedures were harmonized before the study started. Spirometry was systematically performed before the exercise test with a flow volume curve and measurement of forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and the FEV1/FVC ratio (FEV1/FVC), with normalization to Global Lung Function Initiative (GLI) 2012 Z scores. The same investigator coordinator manually calculated the VO2max and the ventilatory anaerobic threshold (VAT) using the V-Slope method. VO2max and VAT values were normalized in a percentage of the predicted VO2max using normal values from Wasserman and Cooper. The investigators considered VO2max below 80% of predicted value as pathologic value and a VAT value below 55 % of predicted VO2max was in favor of muscular deconditioning. All informations from CPET were recorded : heart rate (HR), blood pressure (BP), estimated VO2/HR, VAT, breathing reserves (BR), respiratory rate (RR), The minute ventilation/carbon dioxide production (VE/VCO2 slope), Tidal Volume (VT).

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-17 years old
* Referred to the paediatric cardiopulmonary exercise test (CPET) laboratory of Montpellier University Hospital, France
* Have completed a CPET

  * For cystic fibrosis group:
* To be followed up in the cystic fibrosis center of Montpellier University
* To be referred to our pediatrician CPET laboratory in 2019, or between July and December 2018 if they have not passed a CPET in 201

  • For control group:
* To be referred for non-severe functional symptoms linked to exercise (murmur, palpitation or dyspnea) or for medical sports certificate.
* Having a completely normal check-up, including physical examination, electrocardiogram, echocardiography and spirometry

Exclusion Criteria:

* Patients < 7 ou > 17 years old
* Absolute contraindication for CPET : fever, uncontrolled asthma, respiratory failure, acute myocarditis or pericarditis, uncontrolled arrhythmias causing symptoms or hemodynamic compromise, uncontrolled heart failure, acute pulmonary embolus or pulmonary infarction, and children with mental impairment leading to inability to cooperate
* Parents refuse the use of medical data
* For control group : children with any chronic disease, medical condition (cardiac, neurologic, respiratory, muscular, or renal), medical treatment, requiring any further specialized medical consultation or with any finding at clinical and paraclinical examination (electrocardiogram, echocardiography)

Ages: 7 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children aged 7 to 17 years old recruited in the pediatric CPET laboratory of Montpellier University Hospital, France.
  Cases : children with cystic fibrosis Control : healthy children from a cohort already published (PMID: 29170358)
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen volume by min (VO2 max) assessed by cardiopulmonary exercise test (CPET) | up to 30 oct 2023

SECONDARY OUTCOMES:
Determinants of maximum oxygen volume by min | up to 30 oct 2023
  Assess whether there are determinants that can explain an alteration in vo2max among : anthropometric data, CF-related markers of disease severity including CFTR genotype, pulmonary function test, microbiological data, BHALLA score, pancreatic insufficiency, cystic fibrosis-related diabetes (CFRD), hepatic injury, polyposis, treatments

CONTACTS AND LOCATIONS:
Overall Officials: Johan MOREAU, MD, Principal Investigator — UH Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No